CLINICAL TRIAL: NCT03868553
Title: The Header Burden in Children's and Youth' Football (Soccer)
Brief Title: Header Burden in Football (Soccer)
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: Saarland Header Study
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Header Frequencies, Head Injuries
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Under-10
  Interventions: Other: No intervention
- Under-12
  Interventions: Other: No intervention
- Under-16 female
  Interventions: Other: No intervention
- Under-16 male
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — observational study

SUMMARY:
To assess the realistic magnitude of the header burden in children's and youth' football in eight European countries. In a cross-sectional observational design, one match of 60 different teams in each of the eight European countries were monitored via video recording throughout the second half of the regular season 2017/18 and the first half of the regular season 2018/19. Clubs with (female, male, or mixed) Under-10, Under-12 and female and male Under-16 teams were invited to participate. Header frequencies and types were analysed using standardized heading registration forms. Additionally, head injuries were recorded using standardized head injury registration forms.

ELIGIBILITY:
Inclusion Criteria:

* 1) officially registered in the football association
* 2) regular training participation
* 3) regular participation in official matches

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Football (soccer) playing children and adolescents
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Header frequency | 2018
  Total number of headers and further observations during match play and training sessions

SECONDARY OUTCOMES:
Head injuries | 2018
  Head injuries during match play and training sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University, Saarbrücken, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No
Data were recorded anonymously.